CLINICAL TRIAL: NCT01297647
Title: Incidence of Urinary Tract Infection and Germ Identification After Urodynamic Investigation in Patients With Spinal Cord Injury
Brief Title: Incidence of Urinary Tract Infection After Urodynamic Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Kessler, Executive physician, Balgrist University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 2010-0191/0
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Neurogenic Bladder
Keywords: urinary tract infection; urodynamics; spinal cord injury
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Tract Infections; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal cord injured (Experimental): Patients with neurogenic lower urinary tract infection (Spinal Cord Injury,MS,M. Parkinson)
  Interventions: Procedure: urodynamic examination

INTERVENTIONS:
Procedure: urodynamic examination — Standard urodynamic investigation according to the ICS standard, Good urodynamic practice.Following insertion of 8 F transurethral catheter, retrograde filling of the bladder (20 mL/min) with body warm saline.
  Current recording of pabd. , pves and pdet., subsequently pressure flow study. Additionally imaging with fluoroscopy to detect possible vesico ureteral renal reflux.

SUMMARY:
The purpose of this study is to evaluate the incidence of urinary tract infection after urodynamic investigation and to identify the involved germs.

DETAILED DESCRIPTION:
Patients with neurogenic bladder dysfunction after spinal cord injury need lifelong urologic control examinations with CMG (urodynamic examination). The manipulation may cause urinary tract infections which have to be treated. Patients often noticed an infection after a CMG examination. Aim of this study is the determination of the infection rate and germs. Also should be noticed the pre-interventional infections and differences between the causing germs. Simultaneously the investigators test the reliability of the quicktest for urinary infection. Additionally the investigators will examine the Quality of Life in patients with neurogenic bladder dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurogenic lower urinary tract dysfunction with scheduled urodynamic investigation
* No antibiotic treatment
* Written informed consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Current antibiotic therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary tract infection following urodynamic investigation | 3 days after urodynamic investigation
  every patient receives the urine examination before the urodynamic investigation and hospitalized patients additionally 3 days later and ambulatory patients in case of urinary tract infection

SECONDARY OUTCOMES:
Name and number of identified bacterial species | 30 minutes before examination
Number of hospitalized and number of ambulatory patients with infection of the lower urinary tract | 3 days after examination
Incidence of urinary tract infection before urodynamic investigation | 30 minutes before urodynamic investigation
  every patient receives the urine examination before the urodynamic investigation to detect a potentially urinary tract infection

CONTACTS AND LOCATIONS:
Locations (1):
- Spinal Cord Injury Center & Research, University of Zürich, Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland